CLINICAL TRIAL: NCT05574543
Title: A Randomized, Double-blinded, Placebo-controlled, Phase I/II Study to Evaluate the Safety and Preliminary Efficacy of Single Administration of AGA111 for Lumbar Interbody Fusion in Patients With Degenerative Disc Disease
Brief Title: A Phase I/II Study of AGA111 for Lumbar Interbody Fusion in Patients With Degenerative Disc Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Angitia Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT19001
Record Dates: First submitted 2022-09-30; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.25 mg AGA111 (Experimental): 0.25 mg AGA111 in autologous blood coagulum (ABC) is locally delivered at the intervertebral space.
  Interventions: Drug: AGA111
- 0.5 mg AGA111 (Experimental): 0.5 mg AGA111 in ABC is locally delivered to the participants at the intervertebral space.
  Interventions: Drug: AGA111
- Placebo (Placebo Comparator): Placebo in ABC is locally delivered at the intervertebral space.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGA111 — AGA111 is locally administered in an ABC carrier at the intervertebral space during the lumbar interbody fusion.
  Arms: 0.25 mg AGA111; 0.5 mg AGA111
Drug: Placebo — Placebo is locally administered in an ABC carrier at the intervertebral space during the lumbar interbody fusion.
  Arms: Placebo

SUMMARY:
The objectives of the study are to evaluate the safety and preliminary efficacy of a single administration of AGA111 for lumbar interbody fusion in patients with degenerative disc disease.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, phase 1/2 study to evaluate the safety and preliminary efficacy of single administration of AGA111 for lumbar interbody fusion in patients with degenerative disc disease. A total of 60 participants will be enrolled and randomized to placebo, AGA111 0.25 mg, or AGA111 0.5 mg at 1: 1: 1 ratio. All participants will undergo lumbar interbody fusion and receive study treatment during the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and capable of giving signed informed consent.
2. Male or female, age between 40-80 years.
3. Male or female of childbearing potential must agree to use a highly effective contraception throughout the entire study period, and female subjects must have a negative pregnancy test prior to the randomization.
4. Has degenerative disc disease (DDD) of the lumbosacral(L3-S1) spine that results in back pain, with or without radiating leg pain.
5. Has radiographic evidence (e.g. CT, MRI, x-ray, etc.) of degenerative disc disease.
6. Planning to receive single-level lumbar interbody fusion.
7. Willing and capable of adhering to the protocol and visit schedule.

Exclusion Criteria:

1. Prior surgical procedure at the involved or adjacent spinal levels.
2. Presence or prior history of inflammatory disease of the spine.
3. Presence or prior history of neoplastic disease of the spine.
4. BMI <18.5 or BMI >35.
5. Documented titanium allergy or intolerance.
6. Presence or prior history of malignancy (except for fully resected basal cell carcinoma of the skin).
7. Presence or history of an uncontrolled, unstable, clinically significant medical condition that, in the opinion of the investigator, could jeopardize or compromise the subject's safety or ability to participate in this study.
8. Active local or systemic infection.
9. Female subject who is pregnant or lactating.
10. Serological evidence of positive human immunodeficiency virus (HIV) antibody.
11. HBsAg positive or HBeAg positive, along with positive HBV DNA test.
12. Serological evidence of HCV antibody, along with HCV RNA > lower limit of detection.
13. Known drug or alcohol abuser.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 12 months
  An adverse event (AE) is any untoward medical occurrence in clinical study participant, temporally associated with the use of the investigational product (IP), whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP.
Number of participants who develop anti-drug antibody to AGA111 | Up to 90 days post operation
  Blood samples taken prior to the operation and 5 days, 28 days and 90 days post operation were tested for anti-AGA111 antibodies using an immunoassay method.

SECONDARY OUTCOMES:
Radiographic fusion success | Up to 12 months post operation
  Radiographic fusion success is defined as evidence of continuous bone bridging from the superior to the inferior vertebrae via CT evaluation and no evidence of motion as defined by less than 3mm translational motion and less than 5° in angular motion at the treated level via hyperextension and hyperflexion X-rays.
New Bone formation | Up to 12 months post operation
  New bone formation is defined as the ratio of successful fusion area to the total area in the transverse plane of CT scan.
Oswestry Disability Index (ODI) | Up to 12 months post operation
  The change of point in ODI from baseline.
Pain score through Visual Analogue Scale (VAS) | Up to 12 months post operation
  The change of point in VAS from baseline.
Maximum Concentration (Cmax) of AGA111 | 90 minutes before administration, and 30 minutes, 1 hour, 6 hours, and 24 hours post administration.
  Maximum concentration of AGA111 after dosing.
Time to maximum concentration (Tmax) of AGA111 | 90 minutes before administration, and 30 minutes, 1 hour, 6 hours, and 24 hours post administration.
  Time to maximum concentration of AGA111 after dosing.
Area under the concentration time curve (AUC) | 90 minutes before administration, and 30 minutes, 1 hour, 6 hours, and 24 hours post administration.
  Definite integral of the curve describing the variation of AGA111 in blood as a function of time.

CONTACTS AND LOCATIONS:
Overall Officials: Angitia Medical Director, Study Director — Angitia Medical Director
Locations (6):
- China (6):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No